CLINICAL TRIAL: NCT06122350
Title: The Effect of Earthquake Preparedness Training Given to Mothers With Physically Disabled Children on Psychological Resilience and Earthquake Readiness Levels
Brief Title: Training Given to Mothers With Physically Disabled Children
Acronym: Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Abdullah Adiyaman, Graduate Student, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: YuzuncıYıl
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Earthquake; Physically Disabled
Keywords: Physical Disability; Child; Psychological Resilience; Earthquake; Earthquake preparedness

STUDY DESIGN:
Intervention Model Description: The research was planned as a cross section (pre-test post-test, experimental and control group) randomized controlled study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will be trained within the scope of the Earthquake Preparedness Guide.
  Interventions: Behavioral: Earthquake preparedness training
- Control Group (No Intervention): No intervention will be applied.

INTERVENTIONS:
Behavioral: Earthquake preparedness training — Mothers with physically disabled children will be trained on what to do before, during and after an earthquake within the scope of earthquake preparedness training.
  Arms: Experimental Group

SUMMARY:
Although there are many studies evaluating the effects of earthquakes and earthquakes on humans in our country and in the world, studies evaluating the effects of earthquakes on children with physical disabilities and parents of children with physical disabilities are limited. It is reported that the psychological resilience levels of mothers with disabled children and their level of preparedness for disasters (earthquake, flood, etc.) are low. For this reason, it is important to raise awareness about earthquake preparedness in mothers. This study aims to evaluate the effect of earthquake preparedness training to be given to parents with physically disabled children on the psychological resilience and disaster preparedness levels of mothers.

DETAILED DESCRIPTION:
Earthquakes are recognized as one of the most destructive disasters that cause many people to lose their lives in the world and in Turkey. Due to earthquakes, societies can be exposed to serious economic, social, physical and psychological effects. It has been stated that the most vulnerable members of society are the elderly, children and the disabled. As a matter of fact, it is obvious that the most vulnerable individuals in earthquakes are disabled people with special needs. It was stated that both being a child and being disabled in earthquakes significantly increases vulnerability. In addition, when the studies are examined, it is stated that parents with disabled children are disadvantaged in terms of quality of life, care burden, psychological, economic and social aspects. It has been reported that the disadvantages of parents with physically disabled children increase in earthquakes and they need support in many areas.

Although there are many studies evaluating the effects of earthquakes and earthquakes on humans in our country and in the world, it is seen that studies evaluating the effects of earthquakes on children with physical disabilities and parents of children with physical disabilities are limited. There are studies in which the psychological resilience levels of mothers with disabled children and their readiness levels for disasters (earthquake, flood, etc.) are low. The aim of this study was to evaluate the effect of earthquake preparedness training to be given to parents with physically disabled children on the psychological resilience and disaster preparedness levels of mothers.

ELIGIBILITY:
Inclusion Criteria:

* Having a physically disabled child,
* Literate mothers
* Willing to participate in the study voluntarily,
* The mother who will participate in the study does not have any physical and psychological disorders,
* Mothers who were open to communication were determined as inclusion criteria.

Exclusion Criteria:

* No children with physical disabilities,
* Illiterate,
* Mothers with any physical or psychological illness,
* Mothers who did not want to participate in the study and who were closed to communication were determined as exclusion criteria

Ages: 21 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mothers with Physically Disabled Children
Enrollment: 78 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Psychometric Properties of Adult Resilience Measure (ARM) | 2 monts
  The scale has shown to have good psychometric properties in individuals aged 21 years and above.The four-factor structure of the scale explained 65% of the total variance. The total internal consistency coefficient of the scale was calculated as .94. The test-retest coefficient of the scale was found to be .85. In addition, confirmatory factor analysis results showed that the scale produced good fit values. In conclusion, the results of the study showed that the Adult Resilience Scale and its subscales can be used to measure psychological resilience in adults.
Disaster Preparedness Scale | 2 monts
  The Disaster and Readiness Scale consists of 15 questions and 4 sub-dimensions. The scale explains 59.99 of the total variance. The 4 factors are named as Disaster Physical Protection (DPN), Planning (PP), Disaster Assistance (DAP), Disaster Warning and Signals (DWS) respectively. AFP consists of 7 items with factor loadings ranging from .79 to .40; its mean was 13.76 (X=13.76; SD=4.52, N=1134) and explained 34.47% of the total variance.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Van Yuzuncu Yil Universitesdi, Van
  - Van Yuzuncu Yıl University, Van

IPD SHARING:
Plan to Share IPD: No